CLINICAL TRIAL: NCT01600053
Title: A Phase II Trial of Revlimid® as Consolidation Treatment of Residual Disease in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Revlimid® as Consolidation Treatment Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: interim analysis showed that the trial will not meet the interim endpoint.
Sponsor: Thomas Kipps (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Thomas Kipps, Interim Director, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101955
Record Dates: First submitted 2012-05-09; First posted 2012-05-16 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic; Lymphocytic; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Bronchiolitis Obliterans Syndrome; Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide will be taken orally days 1-21 for up to six 28-day cycles
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide will be taken orally days 1-21 for up to six 28-day cycles (6 cycles = 1 course of Revlimid consolidation). Revlimid will be initiated at 5mg and can be dose escalated at the start of each cycle based on individual patient tolerability to a maximum of 25 mg. The total number of treatment cycles cannot exceed 12 cycles or two courses of six cycles each.
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine whether on course (6 cycles) of consolidation therapy with Revlimid can shrink or slow the growth of Chronic Lymphocytic Leukemia (CLL) in the bone marrow.

DETAILED DESCRIPTION:
CLL is the most prevalent leukemia in the western world and is considered incurable. Standard therapy for CLL is typically in the form of purine analogs, alkylating agents, monoclonal antibodies, or combinations of these drugs. Unfortunately, despite high response rates these treatment strategies are considered palliative and all patients eventually experience disease relapse and with time become less responsive to therapy. Following standard treatment, CLL patients often fail to achieve a complete response, or they have minimal residual disease (MRD) in the marrow and this often correlates with a short time to progression and next therapy.

The National California Institute Working Group and newly updated International Workshop on Chronic Lymphocytic Leukemia Working Group definition of a complete response (CR) in CLL is quite permissive and allows for the persistence of 30% of residual lymphocytes in the marrow. These response criteria were initially developed at a time treatment options for CLL patients were limited and relatively few CRs were obtained. However, therapeutic advances including monoclonal antibodies and stem cell transplant have reduced residual CLL cells to a greater extent than previously possible and necessitated updating of current response criteria to include MRD evaluation and the development of highly sensitive assays that can measure MRD such as multiparametric 4-color flow cytometry, allele-specific PCR, and more convenient investigational assays such as peripheral blood levels of CLLU-1. Regardless, the majority of complete responses achieved following any initial therapy still have detectable residual disease.

Importantly, CLL patients who lack minimal residual disease following treatment consistently demonstrate prolonged progression free survival (PFS) and overall survival (OS) compared with those with persistent MRD. As such, the development of therapeutic strategies that have the potential to eradicate disease after therapy are highly desired. Such consolidation therapies have potential to improve the depth of a remission, prolong PFS, and potentially overall survival in CLL patients. The investigators propose that Revlimid might be one such therapy that can be used as consolidation to eradicate residual disease or improve remissions in patients who have received therapy and that this might lead to a prolonged disease free duration. The investigators hypothesize that Revlimid will be safe and well tolerated in this setting.

The investigators further hypothesize that Revlimid consolidation might be effective in CLL patients at risk of early relapse such as those patients with leukemia cells that use unmutated immunoglobulin heavy chain variable regions. The investigators found that the relative CLLU1 expression level on blood samples mirrored the residual level of CLL cells as determined by 4-color flow cytometry on cells from the aspirated marrow. The investigators hypothesize that monitoring for expression of CLLU1 might provide a reliable means with which to evaluate residual disease in the context of Revlimid consolidation therapy. Previous single agent Revlimid studies have suggested that Revlimid treatment of CLL patients may positively impact immune parameters increasing the relative composition of T-lymphocytes, modulation of cytokines, and can lead to improvement immunoglobulin levels and or the development of leukemia specific antibodies, the investigators hypothesize that similar changes in immune parameters may occur in the context of Revlimid consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia:
* Previously treated patients of any age with a diagnosis of CLL with documented residual disease following therapy, but not meeting an indication for treatment based on current guidelines
* At least 2 months following previous CLL directed therapy
* ECOG performance status of less than or equal to 2 at study entry
* Laboratory test results within these ranges:

  * Platelet count greater than or equal to 50 x 109/L
  * CrCl >.60 ml/min
  * Total bilirubin less than or equal to 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) less than or equal to 2 x ULN
* Females of childbearing must adhere to strict guidelines and have negative pregnancy test prior to enrollment
* Understand and voluntarily sign an informed consent form.
* Age greater than or equal to 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Disease free of prior malignancies for greater than or equal to 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ" of the cervix or breast.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to aspirin may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Known Hepatitis B Ag positive, Hepatitis C positive patients.
* Known HIV positive patients.
* Patients with uncontrolled Autoimmune Hemolytic Anemia (AIHA) or autoimmune thrombocytopenia (ITP)
* Patients with active fungal, bacterial, and/or viral infection
* Patients with known hypersensitivity to Revlimid or thalidomide
* Concurrent use of other anti-cancer agents or treatments
* Patients with history of deep venous thrombus or pulmonary embolism
* Patients who are at increased risk of thrombosis during treatment with Revlimid including those taking concurrent erythropoietin, darbepoetin or high-dose corticosteroids
* Inability to provide informed consent.
* Concurrent malignancy (excluding basal and squamous cell skin cancers).
* Pregnant or breast-feeding females. (Lactating females must agree not to breast feed while taking Revlimid).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Patients with a history of embolic events (e.g. TIA) from arrhythmia or peripheral arterial disease or of recent MI whether or not treated with anti-platelet drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Kipps, M.D., Ph.D., Principal Investigator — University of California Medical Center
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 11
Completed | 0
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — trial will not meet the interim endpoint | 9

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 6
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Eradication of Residual Disease From the Marrow
Time Frame: From date of first dose until then end of 12 cycles of treatment (12 months) or progression of disease, whichever comes first.
Population: This study has been terminated. Interim analysis showed that the trial will not meet the interim endpoint. Data were not collected from the 11 participants before study termination.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

2. Secondary Outcome: Recording of the Occurrence of Adverse Events
Time Frame: From date of first dose until the date of first documented progression or date of death from any cause, whichever came first
Population: This study has been terminated. Interim analysis showed that the trial will not meet the interim endpoint. Please see adverse event listing for additional information.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
participants | 11

ADVERSE EVENTS:
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=11)
cough (General disorders) | 6 (6)
non-cardiac chest pain (General disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 5 (5)
pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
throat pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1)
conjunctivitis (Infections and infestations) | 1 (1)
sinusiitis (Infections and infestations) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 7 (7)
headache (Nervous system disorders) | 4 (4)
fever (General disorders) | 1 (1)
neuropathy (Nervous system disorders) | 4 (4)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 4 (4)
URI (Infections and infestations) | 3 (3)
neutropenia (Blood and lymphatic system disorders) | 9 (10)
hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
anemia (Blood and lymphatic system disorders) | 3 (3)
hyponatremia (Metabolism and nutrition disorders) | 6 (6)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
fatigue (General disorders) | 5 (5)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
colitis (Gastrointestinal disorders) | 1 (1)
rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
small intestine infection (Infections and infestations) | 1 (1)
hypomagnesium (Metabolism and nutrition disorders) | 5 (5)
elevated AST (Investigations) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2)
eye pain (Eye disorders) | 2 (2)
blurred vision (Eye disorders) | 1 (1)
stomach pain (Gastrointestinal disorders) | 1 (1)
elevated ALT (Investigations) | 6 (6)
hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
elevated creatine (Investigations) | 1 (1)
weight loss (Investigations) | 1 (1)
dry eyes (Eye disorders) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
tremors (Nervous system disorders) | 2 (2)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
urinary frequency (Renal and urinary disorders) | 1 (1)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 3 (3)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes